CLINICAL TRIAL: NCT06771908
Title: THE ROLE OF HEXAMIDINE DIISETHIONATE (ZAMIDINE®) 1MG/ML 0.6ML EYE DROPS IN THE PROPHYLAXIS OF SURGERY OFTALMIC
Acronym: ZAMI-PRO
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, RIZZO STANISLAO, Director, Prof, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 7172
Record Dates: First submitted 2025-01-08; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Eye Disease; Conjunctivitis
Keywords: Ophthalmic prophylaxis; Surgery; Ophthalmic Swab
MeSH Terms: conditions — Eye Diseases; Conjunctivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who need ophthalmic surgery: Patients with a history of recurrent conjunctivitis who are scheduled for minor or major ocular surgery.
  Interventions: Diagnostic Test: Conjunctival Swab

INTERVENTIONS:
Diagnostic Test: Conjunctival Swab — CFU/ml by bacterial species before and after prophylaxis.

SUMMARY:
Data will be gathered from patients who report having any kind of recurrent conjunctivitis and who, in accordance with clinical practice, are scheduled to have intravitreal injections, glaucoma surgery, cataract surgery, vitrectomy, combined cataract and vitrectomy, or corneal transplantation.

The data will be obtained using pseudonyms from the patients' medical records and will include the outcomes of swabs and surgeries performed in accordance with clinical practice for the patient's condition.

The following swabs will be taken into consideration for data analysis:

Four days before to surgery, a conjunctival swab is used to check for the presence and load of species that do not make up the typical conjunctival flora (Baseline-T0).

On the day of operation, a conjunctival swab is taken before to entering the recovery room (T1).

Following three minutes of 5% iodopovidone instillation in the eye to be operated on, a conjunctival swab (T2) was used.

Additionally, we will gather follow-up data from the medical record 24 and 30 hours after surgery (at day 34 +/- 7 days).

DETAILED DESCRIPTION:
To determine if Zamidine® reduces ocular surface bacterial flora in surgical prophylaxis.

Secondary goals. To quantify and qualitatively evaluate ocular surface bacterial flora,

* Compare bacterial load before and after surgery with 5% iodopovidone.
* Determine sample endophthalmitis incidence. The study will include patients who are scheduled for intravitreal injections, glaucoma surgery, cataract surgery, vitrectomy, combined cataract and vitrectomy, corneal transplantation, and any type of recurrent conjunctivitis.

Data from patients' medical records will be pseudonymized and contain swabs and operation findings according to clinical practice for their condition.

Following swabs will be analyzed for data:

- a conjunctival swab four days before surgery to detect and quantify non-native organisms.

A conjunctival swab before operation day's recovery room (T1).

- a conjunctival swab (T2) after 3 minutes of 5% iodopovidone in the operative eye.

Follow-up data at 24 and 30 days after surgery (day 34 +- 7 days) will be collected from the medical record.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older, male and female;
2. Patient requiring ophthalmic surgery (intravitreal injections, glaucoma surgery, cataract surgery, vitrectomy, combined cataract and vitrectomy, corneal transplantation) and in need of antiseptic surgical prophylaxis (e.g., Zamidine®)
3. Positive history of recurrent conjunctivitis in the eye requiring surgery.
4. Written informed consent.

Exclusion Criteria:

1. Age < 18 years;
2. Refusal to give informed consent.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Saranno inclusi nello studio i pazienti che devono eseguire qualsiasi intervento di chirurgia oftalmica minore o maggiore con anamnesi positiva di congiuntiviti ricorrenti, secondo pratica clinica e che necessitano di profilassi chirurgica antisettica.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Bacterial species before and after prophylaxis. | 4 days before prophylaxis, the day of surgery before and after povidone-iodine
  CFU/ml by bacterial species before and after prophylaxis.

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Stanislao Rizzo, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Merani R, Hunyor AP. Endophthalmitis following intravitreal anti-vascular endothelial growth factor (VEGF) injection: a comprehensive review. Int J Retina Vitreous. 2015 Jul 21;1:9. doi: 10.1186/s40942-015-0010-y. eCollection 2015. PMID 27847602
- [Background] Speaker MG, Milch FA, Shah MK, Eisner W, Kreiswirth BN. Role of external bacterial flora in the pathogenesis of acute postoperative endophthalmitis. Ophthalmology. 1991 May;98(5):639-49; discussion 650. doi: 10.1016/s0161-6420(91)32239-5. PMID 2062496
- [Background] Peyman A, Hosseini M, Narimani T. Comparison of the Effects of Povidone-Iodine 5%, Polyhexamethylene Biguanide, and Chlorhexidine as a Preoperative Antiseptic in Endophthalmitis Prophylaxis in Patients Undergoing Phacoemulsification Cataract Surgery. Adv Biomed Res. 2020 Apr 22;9:15. doi: 10.4103/abr.abr_155_19. eCollection 2020. PMID 32775308
- [Background] Aragona P, Baudouin C, Benitez Del Castillo JM, Messmer E, Barabino S, Merayo-Lloves J, Brignole-Baudouin F, Inferrera L, Rolando M, Mencucci R, Rescigno M, Bonini S, Labetoulle M. The ocular microbiome and microbiota and their effects on ocular surface pathophysiology and disorders. Surv Ophthalmol. 2021 Nov-Dec;66(6):907-925. doi: 10.1016/j.survophthal.2021.03.010. Epub 2021 Apr 2. PMID 33819460